CLINICAL TRIAL: NCT04594083
Title: A Comparison of Two Different Tactile Stimulus Methods on Reducing Pain
Brief Title: Two Different Tactile Stimulus Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Mürşide Zengin, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/146
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: pain management; child; nursing practice; Intramuscular Injection
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, and experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palm Stimulator (Experimental): The Palm Stimulator was placed in the palm of the child's active hand 20 seconds before the injection. It ensured by researcher that the apparatus was held tightly in the child's palm throughout the procedure. The apparatus was taken back from the child after completing the injection process.
  Interventions: Device: Palm Stimulator
- ShotBlocker (Experimental): ShotBlocker was placed in the ventrogluteal area properly 20 seconds before injection. It was fixed at the injection site until the injection process was completed.
  Interventions: Device: ShotBlocker
- Control (No Intervention): The routine IM injection was applied to the children in the control group.

INTERVENTIONS:
Device: Palm Stimulator — The Palm Stimulator, developed by the present researchers for the first time, is 1.6 cm in diameter, 4 cm in length, and has a cylindrical, non-slippery structure for an easy grip to ensure maximum contact with the palm The Palm Stimulator consists of blunt protrusions that will provide a tactile stimulus on the palm. The blunt protrusions do not penetrate into the skin. The simulator design is based on the gate-control theory, which allows for a reduction in the perceived amount of pain experienced during injection by closing the pain gate in the spinal cord in creating a stimulus on the skin.
  Arms: Palm Stimulator
Device: ShotBlocker — ShotBlocker was placed in the ventrogluteal area properly 20 seconds before injection. It was fixed at the injection site until the injection process was completed.
  Arms: ShotBlocker

SUMMARY:
This study was conducted to evaluate the effects of the ShotBlocker and Palm Stimulator, developed by researchers for reducing pain during intramuscular (IM) injections in children.

DETAILED DESCRIPTION:
Objectives: This study was conducted to evaluate the effects of the ShotBlocker and Palm Stimulator, developed by researchers for reducing pain during intramuscular (IM) injections in children.

Design: The study was conducted via a randomized controlled design. Setting: The study population consisted of children in the seven to 10 age group admitted to the emergency department of a public hospital (Kahta State Hospital) between February 2019 and July 2019 and who received an IM injection as part of the medical treatment.

Interventions: The study data were collected from the children, who were divided into Palm Stimulator, ShotBlocker, and control groups.

Main outcome measures: The children's pre-procedure fear levels were evaluated using the Children's Fear Scale (CFS), and their pain levels during the procedure were evaluated using the Facial Pain Scale-Revised (FPS-R). The children also reported injection-related pain levels using the Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria: children who

* had no diagnosed physical or mental disability or chronic illness;
* had no communication problems;
* received single injection,
* required Ampicillin + Sulbactam group of antibiotics for standardization; and
* received ventrogluteal muscle injection during the study.

Exclusion Criteria:

* Parents who were unable to collaborate in the fear and pain evaluation,
* overweight or underweight children (under the third or above the 97th percentile),
* children with any incision or scar tissue in the injection area,
* children who received a sedative, analgesic, or narcotic drugs (based on expert opinion) six hours before the procedure on the basis of parental statements and medical history

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Children's Fear Scale (CFS) | 5 months
  The Children's Fear Scale (CFS) is a scale used to assess the level of anxiety in children. The scale is a visual measurement tool with scores ranging from 0-4 points. It consists of five facial expressions, ranging from a neutral to a frightened expression, and is suitable for use with children aged 5-10 years (Inan & Inal, 2019; McMurtry, Noel, Chambers, & McGrath, 2011; Özalp Gerçeker, Ayar, Özdemir, & Bektaş, 2018). The evaluation of the Turkish psychometric properties of the scale, which was developed by McMurty et al. for paediatric patients, was conducted by Özalp Gerçeker et al. (2018), and the scale was translated into the Turkish language (Özalp Gerçeker et al., 2018). The CFS has demonstrated good evidence of test-retest (r = 0.76, p < 0.001), and inter-rater (0.51, P < 0.001) reliability, as well as construct validity, (rs ¼ when used with children (McMurtry vd., 2011).
Faces Pain Scale-Revised (FPS-R) | 5 months
  The Faces Pain Scale-Revised (FPS) is a scale used to assess the level of pain in children in the 4-12 age group (Hicks, Von Baeyer, Spafford, Van Korlaar, & Goodenough, 2001). There are facial expressions that show the increasing levels of pain severity from left to right in the scale. Rated according to the severity of pain (between 0-10 points), the leftmost face refers to "no pain", and the rightmost face refers to "too much pain", comprising a total of six facial expressions. The faces exhibit an increase in pain severity to correspond with the scores 0, 2, 4, 6, 8, and 10 from left to right, respectively (Mohamed Mohamed Tork, 2017).
Visual Analog Scale (VAS) | 5 months
  The VAS consists of a horizontal or vertical ruler 10 cm/100 mm in length, with the phrase "no pain" on one end and "the worst pain imaginable" on the other. The child is asked to mark the point on this line that most accurately reflects his/her pain. The distance between the child's mark and the left end of the scale is measured in cm and recorded as "points". It has been suggested that the widely researched scale should be used for children aged seven and older (Çelik & Khorshid, 2015; Sivri Bilgen & Balcı, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Mürşide Zengin, Principal Investigator — Adiyaman University; Emriye Hilal Yayan, Principal Investigator — İnönü University
Locations (1):
- Kahta State Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No